CLINICAL TRIAL: NCT05601544
Title: The Effects of Contact Lenses With UV/HEV-Filter on Visual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6480
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Sphere TEST/CONTROL (Experimental): Eligible subjects who are habitual wearers of soft contact lenses that receive the sphere lenses will be randomized into the sphere TEST/CONTROL sequence.
  Interventions: Device: ACUVUE OASYS 1-Day; Device: ACUVUE OASYS MAX 1-Day
- Sphere CONTROL/TEST (Experimental): Eligible subjects who are habitual wearers of soft contact lenses that receive the sphere lenses will be randomized into the sphere CONTROL/TEST sequence.
  Interventions: Device: ACUVUE OASYS 1-Day; Device: ACUVUE OASYS MAX 1-Day
- Multifocal TEST/CONTROL (Experimental): Eligible subjects who are habitual wearers of soft contact lenses that receive the multifocal lenses will be randomized into the multifocal TEST/CONTROL sequence.
  Interventions: Device: ACUVUE OASYS Multifocal; Device: ACUVUE OASYS MAX 1-Day Multifocal
- Multifocal CONTROL/TEST (Experimental): Eligible subjects who are habitual wearers of soft contact lenses that receive the multifocal lenses will be randomized into the multifocal CONTROL/TEST sequence.
  Interventions: Device: ACUVUE OASYS Multifocal; Device: ACUVUE OASYS MAX 1-Day Multifocal
- Toric TEST/CONTROL (Experimental): Eligible subjects who are habitual wearers of soft contact lenses that receive the toric lenses will be randomized into the toric TEST/CONTROL sequence.
  Interventions: Device: ACUVUE OASYS 1-Day for Astigmatism; Device: senofilcon A based contact lens (toric) with new UV/HEV filter
- Toric CONTROL/TEST (Experimental): Eligible subjects who are habitual wearers of soft contact lenses that receive the toric lenses will be randomized into the toric CONTROL/TEST sequence.
  Interventions: Device: ACUVUE OASYS 1-Day for Astigmatism; Device: senofilcon A based contact lens (toric) with new UV/HEV filter

INTERVENTIONS:
Device: ACUVUE OASYS 1-Day — Sphere CONTROL
  Arms: Sphere CONTROL/TEST; Sphere TEST/CONTROL
Device: ACUVUE OASYS MAX 1-Day — Sphere TEST
  Arms: Sphere CONTROL/TEST; Sphere TEST/CONTROL
Device: ACUVUE OASYS Multifocal — Multifocal CONTROL
  Arms: Multifocal CONTROL/TEST; Multifocal TEST/CONTROL
Device: ACUVUE OASYS MAX 1-Day Multifocal — Multifocal TEST
  Arms: Multifocal CONTROL/TEST; Multifocal TEST/CONTROL
Device: ACUVUE OASYS 1-Day for Astigmatism — Toric CONTROL
  Arms: Toric CONTROL/TEST; Toric TEST/CONTROL
Device: senofilcon A based contact lens (toric) with new UV/HEV filter — Toric TEST
  Arms: Toric CONTROL/TEST; Toric TEST/CONTROL

SUMMARY:
This is a 2-phase, single-site, non-dispensing, randomized, controlled, double-masked, 2x2 crossover study to objectively measure potential benefits of a new UV/HEV filter using psychophysical testing techniques.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 70 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear soft contact lenses (sphere, multifocal, toric) in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.
5. If applicable, those subjects receiving the spherical lenses will need a vertex-corrected distance refraction within the range of -1.00 through -6.00 DS
6. If applicable, those subjects receiving the multifocal lenses will need a vertex-corrected distance refraction within the range of -1.00 through -6.00 DS
7. If applicable, those subjects receiving the toric lenses will need a vertex-corrected distance refraction within the range of -1.50 through -4.00 DS, -0.625 through -1.625 DC, and cylinder axes: 80/90/100, 170/180/10
8. The best corrected, monocular, distance visual acuity must be 20/25 or better in each eye

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. Be currently using any ocular medications or have any ocular infection of any type.
3. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
4. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
5. Be currently wearing lenses in an extended wear modality.
6. Have participated in a contact lens or lens care product clinical trial within 14 days prior to study enrollment.
7. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
8. (Phase 2 only): Have participated in Phase 1 of the study.
9. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
10. Have a history of strabismus or amblyopia.
11. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
12. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- The University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 subjects (only sphere and multifocal subjects) were enrolled into Phase 1 of this study and 0 subjects failed to meet all eligibility criteria. All 21 subjects were dispensed at least 1 study lens and completed Phase 1.
  124 subjects were enrolled into Phase 2. Of those enrolled into Phase 2, 121 subjects were dispensed at least 2 study lenses, while 3 subjects failed to meet all eligibility criteria. 120 subjects completed and 1 subject discontinued from the study during Phase 2.
Groups:
- Senofilcon A (Test) / Senofilcon A (Control) Sphere Strata: Subjects randomized to this sequence are spherical contact lens wearers that received the Test lens during the first period and then received the Control lens during the second period
- Senofilcon A (Control)/ Senofilcon A (Test) Sphere Strata: Subjects randomized to this sequence are spherical contact lens wearers that received the Control lens during the first period and then received the Test lens during the second period
- Senofilcon A (Test) / Senofilcon A (Control) Multifocal Strata: Subjects randomized to this sequence are multifocal contact lens wearers that received the Test lens during the first period and then received the Control lens during the second period
- Senofilcon A (Control) / Senofilcon A (Test) Multifocal Strata: Subjects randomized to this sequence are multifocal contact lens wearers that received the Control lens during the first period and then received the Test lens during the second period
- Senofilcon A (Test) / Senofilcon A (Control) Toric Strata: Subjects randomized to this sequence are toric contact lens wearers that received the Test lens during the first period and then received the Control lens during the second period
- Senofilcon A (Control) / Senofilcon A (Control) Toric Strata: Subjects randomized to this sequence are toric contact lens wearers that received the Control lens during the first period and then received the Control lens during the second period
Period: Phase 1 Period 1
Arm/Group | Senofilcon A (Test) / Senofilcon A (Control) Sphere Strata | Senofilcon A (Control)/ Senofilcon A (Test) Sphere Strata | Senofilcon A (Test) / Senofilcon A (Control) Multifocal Strata | Senofilcon A (Control) / Senofilcon A (Test) Multifocal Strata | Senofilcon A (Test) / Senofilcon A (Control) Toric Strata | Senofilcon A (Control) / Senofilcon A (Control) Toric Strata
Started | 5 | 6 | 5 | 5 | 0 | 0
Completed | 5 | 6 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1 Period 2
Arm/Group | Senofilcon A (Test) / Senofilcon A (Control) Sphere Strata | Senofilcon A (Control)/ Senofilcon A (Test) Sphere Strata | Senofilcon A (Test) / Senofilcon A (Control) Multifocal Strata | Senofilcon A (Control) / Senofilcon A (Test) Multifocal Strata | Senofilcon A (Test) / Senofilcon A (Control) Toric Strata | Senofilcon A (Control) / Senofilcon A (Control) Toric Strata
Started | 5 | 6 | 5 | 5 | 0 | 0
Completed | 5 | 6 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 Period 1
Arm/Group | Senofilcon A (Test) / Senofilcon A (Control) Sphere Strata | Senofilcon A (Control)/ Senofilcon A (Test) Sphere Strata | Senofilcon A (Test) / Senofilcon A (Control) Multifocal Strata | Senofilcon A (Control) / Senofilcon A (Test) Multifocal Strata | Senofilcon A (Test) / Senofilcon A (Control) Toric Strata | Senofilcon A (Control) / Senofilcon A (Control) Toric Strata
Started | 20 | 21 | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20 | 20 | 20
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Phase 2 Period 2
Arm/Group | Senofilcon A (Test) / Senofilcon A (Control) Sphere Strata | Senofilcon A (Control)/ Senofilcon A (Test) Sphere Strata | Senofilcon A (Test) / Senofilcon A (Control) Multifocal Strata | Senofilcon A (Control) / Senofilcon A (Test) Multifocal Strata | Senofilcon A (Test) / Senofilcon A (Control) Toric Strata | Senofilcon A (Control) / Senofilcon A (Control) Toric Strata
Started | 20 | 20 | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sphere Strata - Phase 1; Sphere Strata - Phase2: Subjects who are spherical contact lens wearers
- Multifocal Strata - Phase 1; Multifocal Strata - Phase 2: Subjects who are multifocal contact lens wearers
- Toric Strata - Phase 2: Subjects who are toric contact lens wearers
- Total: Total of all reporting groups
Arm/Group | Sphere Strata - Phase 1 | Multifocal Strata - Phase 1 | Sphere Strata - Phase2 | Multifocal Strata - Phase 2 | Toric Strata - Phase 2 | Total
Number analyzed (Participants) | 11 | 10 | 41 | 40 | 40 | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All subjects dispensed a study lens in Phase 1
  Years | 23.4 (3.04) | 50.9 (9.88) | 25.8 (6.49) | 51.0 (7.08) | 24.9 (5.28) | 36.5 (15.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 29 | 37 | 30 | 114
  Male | 1 | 2 | 12 | 3 | 10 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 6 | 0 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 5 | 4 | 14
  White | 11 | 7 | 32 | 34 | 33 | 117
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 41 | 40 | 40 | 142

OUTCOME MEASURES:

1. Primary Outcome: Visual Range at Phase 1
Description: Visual range is defined as the log relative energy of simulated haze needed to obscure an otherwise high contrast grating target. Better visual range is indicated by a higher log-relative energy (LRE) of simulated haze (more haze) to obscure an otherwise highly visible target.
Time Frame: Approximately 15 minutes post lens fitting
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from the study or deviation from the protocol.
Measure: Mean (Standard Deviation); unit: log relative energy level
Groups:
- Senofilcon A (Test) Sphere Strata - Phase 1: Spherical subjects that wore the senofilcon A (Test) lens in either the first or second period in Phase 1 of the study.
- Senofilcon A (Control) Sphere Strata - Phase 1: Spherical subjects that wore the senofilcon A (Control) lens in either the first or second period in Phase 1 of the study
- Senofilcon A (Test) Multifocal Strata - Phase 1: Multifocal subjects that wore the senofilcon A (Test) lens in either the first or second period in Phase 1 of the study
- Senofilcon A (Control) Multifocal Strata - Phase 1: Multifocal subjects that wore the senofilcon A (Control) lens in either the first or second period in Phase 1 of the study
Arm/Group | Senofilcon A (Test) Sphere Strata - Phase 1 | Senofilcon A (Control) Sphere Strata - Phase 1 | Senofilcon A (Test) Multifocal Strata - Phase 1 | Senofilcon A (Control) Multifocal Strata - Phase 1
Number analyzed (Participants) | 11 | 11 | 10 | 10
log relative energy level | 3.232 (0.1658) | 3.049 (0.2101) | 3.287 (0.1824) | 3.167 (0.1072)

2. Primary Outcome: Visual Range at Phase 2
Description: as for outcome 1
Time Frame: Approximately 15 minutes post lens fitting
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from the study or deviation from the protocol. Based on the pre-specified primary analyses for Phase 2, the primary hypothesis testing was performed for Sphere and Multifocal strata only.
Measure: Mean (Standard Deviation); unit: log relative energy level
Groups:
- Senofilcon A (Test) Sphere Strata - Phase 2: Spherical subjects that wore the senofilcon A (Test) lens in either the first or second period in Phase 2 of the study.
- Senofilcon A (Control) Sphere Strata - Phase 2: Spherical subjects that wore the senofilcon A (Control) lens in either the first or second period in Phase 2 of the study
- Senofilcon A (Test) Multifocal Strata - Phase 2: Multifocal subjects that wore the senofilcon A (Test) lens in either the first or second period in Phase 2 of the study
- Senofilcon A (Control) Multifocal Strata - Phase 2: Multifocal subjects that wore the senofilcon A (Control) lens in either the first or second period in Phase 2 of the study
Arm/Group | Senofilcon A (Test) Sphere Strata - Phase 2 | Senofilcon A (Control) Sphere Strata - Phase 2 | Senofilcon A (Test) Multifocal Strata - Phase 2 | Senofilcon A (Control) Multifocal Strata - Phase 2
Number analyzed (Participants) | 40 | 41 | 40 | 40
log relative energy level | 3.377 (0.1489) | 3.156 (0.1181) | 3.181 (0.1649) | 3.020 (0.1412)
Statistical Analysis 1: Comparison: Senofilcon A (Test) Sphere Strata - Phase 2 vs Senofilcon A (Control) Sphere Strata - Phase 2; It was calculated that 41 (for the Multifocal strata) and 6 (for the Sphere strata) participants in each vision group randomized in a 1:1 fashion between the two sequences would have at least a power of 90% (for the Multifocal strata) and a power of 94% (for the Sphere strata) to detect a statistical superiority with respect to visual range; Test type: Superiority; p < .0001, Mixed Model Analysis — 1-sided p-value was calculated using one-sided type 1 error of 0.025; the Kenward and Roger method was used for the calculation of the denominator degrees of freedom; Least-squares Mean difference = 0.22, 95% CI 2-sided [0.19 to 0.25], Standard Error of Mean 0.016 — Least-squares mean difference was calculated as Test minus Control
Statistical Analysis 2: Comparison: Senofilcon A (Test) Multifocal Strata - Phase 2 vs Senofilcon A (Control) Multifocal Strata - Phase 2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < .0001, Mixed Model Analysis — 1-sided p-value was calculated using one-sided type 1 error of 0.025; the Kenward and Roger method was used for the calculation of the denominator degrees of freedom; Least-squares Mean difference = 0.16, 95% CI 2-sided [0.14 to 0.18], Standard Error of Mean 0.011 — Least-squares mean difference was calculated as Test minus Control

3. Primary Outcome: Motion Detection at Phase 1
Description: Motion detection is defined as the distance needed (in mm) to determine that a test light has moved from a standard position. Better motion detection is indicated by a smaller distance needed to detect that movement has occurred.
Time Frame: Approximately 15 minutes post lens fitting
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from the study or deviation from the protocol. Subject were analyzed per planned randomized treatment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Senofilcon A (Test) Sphere Strata - Phase 1 | Senofilcon A (Control) Sphere Strata - Phase 1 | Senofilcon A (Test) Multifocal Strata - Phase 1 | Senofilcon A (Control) Multifocal Strata - Phase 1
Number analyzed (Participants) | 11 | 11 | 10 | 10
mm | 1.725 (1.3575) | 2.881 (1.9824) | 3.229 (2.3248) | 2.716 (3.1286)

4. Primary Outcome: Brightness Perception at Phase 1
Description: Brightness perception is defined as the log- relative energy needed to match a standard stimulus to a natural scene, across 10 different projected scenes. The perception of brighter image is indicated by a higher log-relative energy (LRE) needed to match the initially dim standard to the target.
Time Frame: Approximately 15 minutes post lens fitting
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log relative energy
Arm/Group | Senofilcon A (Test) Sphere Strata - Phase 1 | Senofilcon A (Control) Sphere Strata - Phase 1 | Senofilcon A (Test) Multifocal Strata - Phase 1 | Senofilcon A (Control) Multifocal Strata - Phase 1
Number analyzed (Participants) | 11 | 11 | 10 | 10
log relative energy | 1.109 (0.0909) | 1.081 (0.1494) | 1.101 (0.1388) | 1.041 (0.2222)

5. Secondary Outcome: Motion Detection at Phase 2
Description: as for outcome 3
Time Frame: Approximately 15 minutes post lens fitting
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from the study or deviation from the protocol. Subject were analyzed per planned randomized treatment. Based on the pre-specified primary analyses for Phase 2, the primary hypothesis testing was performed for Sphere and Multifocal strata only.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Senofilcon A (Test) Sphere Strata - Phase 2 | Senofilcon A (Control) Sphere Strata - Phase 2 | Senofilcon A (Test) Multifocal Strata - Phase 2 | Senofilcon A (Control) Multifocal Strata - Phase 2
Number analyzed (Participants) | 40 | 41 | 39 | 39
mm | 3.894 (2.6800) | 4.288 (2.9575) | 3.499 (2.4146) | 3.3376 (2.3750)
Statistical Analysis 1: Comparison: Senofilcon A (Test) Sphere Strata - Phase 2 vs Senofilcon A (Control) Sphere Strata - Phase 2; It was calculated that 16 participants in each group randomized in a 1:1 fashion between the two sequences would have at least 92% power to detect a statistical superiority with respect to motion detection; Test type: Superiority; p = 0.0465, Mixed Model Analysis — 1-sided p-value was calculated using one-sided type 1 error of 0.0083; the Kenward and Roger method was used for the calculation of the denominator degrees of freedom; Median Ratio = 0.83, 98.33% CI 2-sided [0.64 to 1.09] — Median Ratio was calculated as test over control

6. Secondary Outcome: Brightness Perception at Phase 2
Description: as for outcome 4
Time Frame: Approximately 15 minutes post lens fitting
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: log relative energy
Arm/Group | Senofilcon A (Test) Sphere Strata - Phase 2 | Senofilcon A (Control) Sphere Strata - Phase 2 | Senofilcon A (Test) Multifocal Strata - Phase 2 | Senofilcon A (Control) Multifocal Strata - Phase 2
Number analyzed (Participants) | 40 | 40 | 40 | 40
log relative energy | 1.356 (0.0670) | 1.222 (0.0615) | 1.360 (0.0832) | 1.219 (0.0843)
Statistical Analysis 1: Comparison: Senofilcon A (Test) Multifocal Strata - Phase 2 vs Senofilcon A (Control) Multifocal Strata - Phase 2; It was calculated that 29 participants in each group randomized in a 1:1 fashion between the two sequences would have at least 91% power to detect a statistical superiority with respect to motion detection; Test type: Superiority; p < .0001, Mixed Model Analysis — 1-sided p-value was calculated using one-sided type 1 error of 0.0083; the Kenward and Roger method was used for the calculation of the denominator degrees of freedom; Least-square Mean Difference = 0.14, 98.33% CI 2-sided [0.112 to 0.170] — Least-square Mean difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Time Frame: Throughout the duration of the study (Phase 1 and Phase 2); approximately 1 month per subject.
Description: All subjects dispensed at least 1 study lens during either Phase 1 or Phase 2 of the study.
Groups:
- Senofilcon A (Control) Multifocal Strata - Phase 2: Multifocal subjects that wore the senofilcon A (Test) lens in either the first or second period in Phase 2 of the study.
- Senofilcon A (Test) Toric Strata - Phase 2: Toric subjects that wore the senofilcon A (Test) lens in either the first or second period in Phase 2 of the study.
- Senofilcon A (Control) Toric Strata - Phase 2: Toric subjects that wore the senofilcon A (Control) lens in either the first or second period in Phase 2 of the study.
Arm/Group | Senofilcon A (Test) Sphere Strata - Phase 1 | Senofilcon A (Control) Sphere Strata - Phase 1 | Senofilcon A (Test) Multifocal Strata - Phase 1 | Senofilcon A (Control) Multifocal Strata - Phase 1 | Senofilcon A (Test) Sphere Strata - Phase 2 | Senofilcon A (Control) Sphere Strata - Phase 2 | Senofilcon A (Test) Multifocal Strata - Phase 2 | Senofilcon A (Control) Multifocal Strata - Phase 2 | Senofilcon A (Test) Toric Strata - Phase 2 | Senofilcon A (Control) Toric Strata - Phase 2
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/10 | 0/40 | 0/41 | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/10 | 0/40 | 0/41 | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10 | 0/10 | 0/40 | 0/41 | 0/40 | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT05601544/Prot_SAP_000.pdf